CLINICAL TRIAL: NCT06564870
Title: Retrospective Observational Study of the Efficacy and Safety of DURVALUMAB Maintenance Therapy in Patients With Stage III Non-Small Cell Lung Cancer (DURVABREIZH)
Brief Title: Efficacy and Safety Study of DURVALUMAB Maintenance in Patients With Stage III Non-Small Cell Lung Cancer
Acronym: DURVABREIZH
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DURVABREIZH - 29BRC21.0199
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Bronchial Cancer
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the real-life efficacy of durvalumab treatment in consolidation after radio-chemotherapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) such as anti-PD-1/PD-L1 have revolutionized the field of immuno-oncology, inducing significant and durable responses in patients with all types of tumor, and in particular advanced stage (II-IV) non-small cell lung cancer (NSCLC). The use of durvalumab in consolidation, after radiochemotherapy, in locally advanced NSCLC has significantly improved progression-free survival and overall survival (see PACIFIC trial). Durvalumab now has marketing authorization for this indication, in cases of PD-L1≥1% overexpression on tumor cells.

However, 50% of patients experience tumor progression at 1 year, and there is currently no biomarker (clinical, biological or radiological) predictive of tumor response to durvalumab in consolidation.

Elucidating the determinants of response and resistance to treatment, as well as predicting severe immune-mediated adverse events, are essential to improving patient outcomes and developing new therapeutic strategies

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable locally advanced non-small-cell lung cancer (stages II, IIIA, IIIB and IIIC) responding to or stable after concomitant or sequential platinum-based radiochemotherapy and having received durvalumab consolidation therapy
* Minimum radiotherapy dose of 54 Gy to 66 Gy
* Age greater than or equal to 18 years
* WHO 0-1
* Non-opposition of living patients formulated

Exclusion Criteria:

* Age < 18 years.
* Refusal to participate
* Patients under legal protection (curatorship, guardianship, etc.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable locally advanced non-small cell lung cancer (stages IIIA, IIIB and IIIC) who have responded to or are stable after concurrent or sequential platinum-based radiochemotherapy and have received maintenance durvalumab therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Real-life efficacy of durvalumab treatment in maintenance after chemoradiotherapy. | 1 year
  progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement